CLINICAL TRIAL: NCT05583084
Title: Sex-unique Disparities in Survival and Resuscitation After Out-of-hospital Cardiac Arrest - a Danish Analysis
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Eleonora Casarini, Fellow researcher and medical student, Prehospital Center, Region Zealand
Other Study IDs: ohcagd2022
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: sex differences; ohca; women; SIR; CPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Contact Tracing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Investigation

SUMMARY:
The goal of this observational study is to investigate characteristics in out-of-hospital cardiac arrests (OHCA) related to sex differences.

The main questions it aims to answer are:

* are there possible differences in help provision by bystanders, cardiopulmonary resuscitation (CPR), pre-hospital treatment by emergency medical services (EMS)?
* are there differences in the presence of shockable initial rhythm (SIR) and survival rates after OHCA at successive stages of treatment? Researchers will compare all emergency medical services treated resuscitations in Denmark between 2016 and 2021 to see if there are possible differences between sexes.

DETAILED DESCRIPTION:
This analysis will be based on data from the national electronic based Danish OHCA registry. Data on OHCAs with resuscitative attempts in Denmark have been collected in the electronic based Danish Medical Service report system since 2016. The registry covers detailed data including the EMS report, executive entries, and advanced text searches of prehospital charts. All cases go through an elaborate validation process where all identified events are read through manually by an external verification team. This ensures high quality of data, collected according to the Utstein recommendations, throughout the approximately 5400 cases of OHCA in Denmark annually. During this verification process, supplementary sources of data are linked to each OHCA, among others information about survival, localization, initiation of bystander CPR and EMS personnel operation.

ELIGIBILITY:
Inclusion Criteria:

- All emergency medical services treated resuscitations in Denmark between 2016 and 2021

Exclusion Criteria:

- Patients that are found dead at emergency medical service arrival, with sure death indicators such as rigor mortis or livores.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All emergency medical services treated resuscitations in Denmark between 2016 and 2021 registered in the national electronic based Danish OHCA registry
Sampling Method: Non-Probability Sample
Enrollment: 27000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
30-days survival | 30 days from OHCA
  Records on survival after 30 days from cardiac arrest

SECONDARY OUTCOMES:
Cardiopulmonary Resuscitation (CPR) | 2016-2021
  Whether or not CPR was performed on the patient
Presence of shockable initial rhythm (SIR) | 2016-2021
  Whether or not a schockable intial rhythm was recorded
Return of spontaneous circulation (ROSC) at any time | 2016-2021
  Whether or not there was return of spontaneous circulation at any time

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT05583084/Prot_000.pdf